CLINICAL TRIAL: NCT03600233
Title: A Phase II, Open-label Study of CVM-1118 Administered Orally to Patients With Advanced Neuroendocrine Tumors
Brief Title: Study of CVM-1118 for Patients With Advanced Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-005
Record Dates: First submitted 2018-06-07; First posted 2018-07-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Tumors; Pancreatic Neuroendocrine Tumor; Gastro-enteropancreatic Neuroendocrine Tumor; Lung Neuroendocrine Neoplasm; Neuroendocrine Carcinoma
Keywords: Oncology; Neuroendocrine Tumors; NET; Vasculogenic mimicry
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell; Gastro-enteropancreatic neuroendocrine tumor; Carcinoma, Neuroendocrine; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVM-1118 (Experimental): CVM-1118 200mg or 300mg Bis In Die (BID) daily/ Cycle (28 days per cycle)
  Interventions: Drug: CVM-1118

INTERVENTIONS:
Drug: CVM-1118 — Patients will initially receive CVM-1118 orally twice daily at 200 mg per dose (400 mg total daily dose).
  Patients who tolerate this dose for at least 2 Cycles will have the option of increasing the dose of CVM-1118 to 300 mg BID (600 mg total daily dose) if specific criteria are met.
  Other Names: TRX-818

SUMMARY:
CVM-1118 (TRX-818) is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by TaiRx, Inc. CVM-1118 is a potent anti-cancer agent in numerous human cancer cell lines. The safety of administrating CVM-1118 on human is evaluated from the phase 1 study. The objectives of the phase 2 study is to further investigate the efficacy of CVM-1118 for patients with advanced neuroendocrine tumors.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a group of uncommon heterogeneous malignancies originating from neuroendocrine cells localized throughout the body. Approximately 50% of patients with NETs would have metastatic cancer, where 65% of patients with metastatic cancer would result in mortality within 5 years of diagnosis.

The current treatments of NETs do not follow single discipline and the effective agents are largely still under clinical investigations. Apparent formation of vasculogenic mimicry (VM) has been reported in at least two types of NETs. Moreover, VM has been found as part of multiple microvascular alterations in mouse models of pancreatic neuroendocrine tumors.

Wih the high potential of inhibiting VM formation, CVM-1118 is considered to have therapeutic potentials in treating NET tumors.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet ALL of the following criteria:

1. [Tumor eligibility] Histologically or cytologically confirmed advanced (unresectable and/or metastatic) neuroendocrine tumors that are well-differentiated, low or intermediate grade (WHO Grade 1 or 2) of pancreatic or gastrointestinal, or low/ intermediate grade of lung origin, that are refractory to standard of care therapy, or for whom no standard of care therapy is available.
2. Patients must have measurable or evaluable disease as per RECIST criteria v1.1. Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy.
3. Patients must have documented progressive disease within 6 months prior enrollment after prior therapy.
4. Patients who are on therapy with a somatostatin analog are eligible but progressive disease must be demonstrated subsequent to establishment for at least 3 months of a stable dose.
5. Male or female, 20 years of age or older.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Resolution of all acute toxic effects of prior therapy or surgical procedures to Grade 1 (except alopecia).
8. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≦ 3 x upper limit of normal (ULN), or AST and ALT ≦ 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≦ 1.5 x ULN (except for patients with documented Gilbert's syndrome)
   * Absolute neutrophil count (ANC) ≧ 1500/µL
   * Platelets ≧ 90,000/µL
   * Hemoglobin ≧ 9.0 g/dL
   * Serum creatinine ≦ 2.0 x ULN or creatinine clearance of ≧ 50 mL/min
9. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

Patients eligible for this study must not meet ANY of the following criteria:

1. Poorly differentiated neuroendocrine carcinoma, or high grade neuroendocrine tumor.
2. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
3. Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of starting study treatment.
4. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
5. Current treatment on another clinical trial.
6. Patients who are using other investigational agents or who had received investigational drugs within 4 weeks prior to study enrollment.
7. Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
8. Any of the following within the 12 months prior to starting study treatment:

   myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and sponsor, the 6-month post-event-free period for a patient with a pulmonary embolus can be waived if due to advanced cancer. Appropriate treatment with anticoagulants is permitted.
9. Hypertension that cannot be controlled by medications (> 160/100 mmHg despite optimal medical therapy).
10. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
11. Known history of human immunodeficiency virus (HIV) seropositivity and/or is receiving anti-retroviral therapy.
12. Hepatitis B virus (HBV) or hepatitis C virus (HCV) with evidence of chronic active disease or receiving/requiring antiviral therapy.
13. History of receiving organ transplantation or immune disorders that require continuous immunosuppressant agent therapy.
14. Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal or must agree to the use of effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the Investigator or a designated associate.
15. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or Sponsor, excess risk associated with study participation or study drug administration, which would make the patient inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time-to progression-free survival (PFS) | 12 months after the last patient enrolled
  Measure the Time-to PFS or death to any cause. The tumor assessment will be performed every 12 weeks until documented disease progression, death, or date of follow-up.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months after the last patient enrolled
  ORR is defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR), based on the investigator's assessment as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1.
Disease control rate (DCR) | up to 12 months after the last patient enrolled
  DCR is defined as the proportion of patients with a best overall response of CR, PR, or Stable Disease (SD), based on the investigator's assessment per RECIST criteria v1.1.
Duration of overall response (DoR) | up to 12 months after the last patient enrolled
  DoR is measured only for the responder subset: patients with confirmed CR or PR based on the investigator's assessment. It is the elapsed time between the date of first documented response and the following date of event defined as the first documented disease progression or death due to underlying cancer, per RECIST criteria v1.1.
Time-to progression (TTP) | up to 12 months after the last patient enrolled
  TTP is defined as the duration of time from initiation of study medication to first documentation of tumor progression.
Time-to overall survival (OS) | up to 12 months after the last patient enrolled
  OS is defined as the duration of time from initiation of study medication to death due to any cause.
Number of participants with treatment-related adverse events (AEs) as assessed by CTCAE v4.03 | During the course of the trial or within 28 days following termination from the trial
  Assessment of adverse events will based on the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE].
Number of Participants With Abnormal baseline and out-of range Hematology Count by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Number of Participants With Abnormal Laboratory Values_Assessed the baseline and out-of range urinalysis test by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided. A list of all laboratory normal ranges will also be provided.
Number of Participants With Abnormal Laboratory Values_Assessed the baseline and out-of range coagulation test by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Normal range of PT/PTT will be provided. Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal laboratory values would be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ body temperature by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ blood pressure by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ heart rate by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Number of Participants With Abnormal Vital Sign_Assessed the baseline and out-of-range vital signs_ respiratory rate by CTCAE v4.03 | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  Values with CTCAE v4.03 Grade ≧ 3 will be identified with flags. A final outcome result with the number of participants with abnormal vital sign would be provided. Normal ranges will also be provided.
Abnormalities in electrocardiography (ECG) | From baseline of screening up to end of treatment or withdraw, an average of 12 months
  a 12-lead (with a 10-second rhythm strip) tracing, with a capacity to calculate the standard intervals automatically, will be used.
Maximum Plasma Concentration [Cmax] of CVM-1118 and its metabolite CVM-1125 after CVM-1118 dosing | Cycle 1 and Cycle 2 (each cycle is 28 days)
  PK parameters will be calculated for CVM-1118 and its metabolite CVM-1125 during this study.
Area Under the Curve [AUC] of CVM-1118 and its metabolite CVM-1125 after CVM-1118 dosing | Cycle 1 and Cycle 2 (each cycle is 28 days)
  PK parameters will be calculated for CVM-1118 and its metabolite CVM-1125 during this study.
Pharmacodynamics analysis for the relationship of Cmax and PFS | Cycle 1 and Cycle 2 (each cycle is 28 days)
  The correlations of PK parameter, Cmax and key efficacy endpoint will be evaluated in this study.
Pharmacodynamics analysis for the relationship of AUC and PFS | Cycle 1 and Cycle 2 (each cycle is 28 days)
  The correlations of PK parameter, AUC and key efficacy endpoint will be evaluated in this study.
Pharmacodynamics analysis for the relationship of AUC and AE | Cycle 1 and Cycle 2 (each cycle is 28 days)
  The correlations of PK parameter, AUC and key safety endpoint will be evaluated in this study.
Pharmacodynamics analysis for the relationship of Cmax and AE | Cycle 1 and Cycle 2 (each cycle is 28 days)
  The correlations of PK parameter, Cmax and key safety endpoint will be evaluated in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, Principal Investigator — National Cheng Kung University Hospital,Taiwan
Locations (8):
- Taiwan (8):
  - Chang Gung Memorial Hospital, KaoHsiung, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, LinKou, Taoyuan